CLINICAL TRIAL: NCT04123314
Title: Pilot Study of Serotonin 2A Receptor (5-HT2A) Agonist Psilocybin for Depression in Patients With Mild Cognitive Impairment or Early Alzheimer's Disease
Brief Title: Psilocybin for Depression in People With Mild Cognitive Impairment or Early Alzheimer's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Council On Spiritual Practices (Unknown); Heffter Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00175915
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Depressive Symptoms; Depression; Alzheimer Disease; Mild Cognitive Impairment
Keywords: Psilocybin; Hallucinogen; Psychedelic
MeSH Terms: conditions — Depression; Alzheimer Disease; Cognitive Dysfunction | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): Participants will complete an 8-week course of study treatment including weekly psychological support and two moderate to high dose psilocybin administrations in weeks 4 and 6.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Dosing at the first session will be 15 mg/70 kg. For the second session participants will either remain at the initial dose, or increase to 25 mg/70 kg at the discretion of the study team.

SUMMARY:
This open-label pilot study examines whether the hallucinogenic drug, psilocybin, given under supportive conditions, is safe and effective for depression in people with Mild Cognitive Impairment (MCI) or early Alzheimer's Disease (AD). This study will also assess whether psilocybin may improve quality of life in those individuals.

DETAILED DESCRIPTION:
This is a pilot study evaluating the potential efficacy of psilocybin to produce improvement in depression compared to pre-treatment in people with Mild Cognitive Impairment (MCI) or early Alzheimer's Disease (AD) and clinically significant symptoms of depression. The study will be an open-label trial in a sample of up to 20 treatment-seeking participants with a diagnosis of MCI or early AD. Participants will complete an 8-week course of study treatment including two psilocybin sessions (15 mg/70 kg in week 4 and 15 or 25 mg/70 kg in week 6), with follow-up assessments up to 6 months after the final psilocybin session. The study will assess changes in depressed mood at 1 week after the second psilocybin session compared to pre-treatment, and quality of life in participants from pre- to post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must meet either A) Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) criteria for Mild Neurocognitive Disorder due to AD or Major Neurocognitive Disorder due to AD with Mild severity (including probable), or B) meet criteria for MCI including a subjective memory complaint relative to previous functioning and confirmed by Clinical Dementia Rating (CDR) Memory score at screening of >0.5
* Have Mini-Mental State Examination scores >18
* Have a Montreal Cognitive Assessment score <26.
* Have Cornell Scale for Depression in Dementia (CSDD) patient score >/= 6, or Geriatric Depression Scale-Short Form score ≥ 5, indicating at minimum a mild to moderate degree of distress.
* Acetylcholinesterase inhibitors are allowed so long as the dose has been stable for > 6 weeks.
* Concurrent pharmacotherapy with selective serotonin reuptake inhibitors (SSRI), serotonin and norepinephrine reuptake inhibitors (SNRI), and/or bupropion is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening. Allowable bupropion doses for participants will be ≤300mg/day.
* Have a close friend or family member willing and able to serve the role of community observer / informant for data collection procedures

Exclusion Criteria:

* Individuals 86 years of age or older will be excluded.
* Currently taking antipsychotics, monoamine oxidase (MAO) inhibitors, or antidepressant medications other than SSRIs, SNRIs, or bupropion. Allowable bupropion doses for participants will be ≤300mg/day.
* Long-acting opioid pain medications (e.g. oxycodone sustained release, morphine sustained release - which are usually taken at 12 hour intervals) will be allowed if the last dose occurred at least 2 hours before psilocybin administration and the next dose was not scheduled until at least 8 hours after psilocybin administration.
* Participants must agree not to take sildenafil, tadalafil, or similar medications within 72 hours of each psilocybin administration, as these medications may potentiate hypotensive reactions to psilocybin
* Cardiovascular conditions: angina, a clinically significant ECG abnormality (e.g. atrial fibrillation or heart-rate corrected QT interval (QTc) >450msec), Transient Ischemic Attack (TIA) in the last 6 months, stroke, artificial heart valves, or uncontrolled hypertension with resting blood pressure systolic >150 or diastolic >95
* Minimum acceptable heartrate at screening is 50 bpm unless the individual is cleared for participation by a cardiologist, in accord with the American College of Cardiology's 2018 guidelines for bradycardia
* Seizure disorder
* Insulin dependent diabetes mellitus
* Renal disease (creatinine clearance < 40 ml/min using the Cockcroft and Gault equation)
* Baseline liver enzyme elevation >2x the upper limit of normal
* Current or past history of meeting DSM-5 criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I Disorder
* Family (i.e., 1st degree relative) history of Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I Disorder
* Past-year hallucinogen use.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cornell Scale for Depression in Dementia (CSDD) score | Baseline and 1 week after second psilocybin session
  The Cornell Scale for Depression in Dementia (CSDD) is administered via patient and informant interviews to assess the presence and severity of depressive mood and behavioral symptoms during the past week. Has 19 items, each scored from 0 to 2 with higher scores indicating severe symptom.Total score range from 0 to 38.

SECONDARY OUTCOMES:
Change in Quality of Life Alzheimer's Disease (QOL-AD) scale score | Baseline and 2 weeks after second psilocybin session
  The Quality of Life Alzheimer's Disease (QOL-AD) scale is a 13-item measure administered via patient and informant interviews to assess overall mood, physical and cognitive function, and quality of relationships in people with Alzheimer's Disease. Each item is scored 1 to 4, with higher score indicating better quality of life. Total score range from 13 to 52.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Garcia-Romeu, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No